CLINICAL TRIAL: NCT01870999
Title: An Open-label Parallel Arm Multiple Dose Tolerability, Pharmacokinetics and Safety Study in Adult Patients With Schizophrenia Following Administration of Aripiprazole IM Depot Formulation Once Every Four Weeks
Brief Title: A Multiple Dose Safety, Tolerability and Pharmacokinetics Study in Adult Patients With Schizophrenia Following Administration of Aripiprazole IM Depot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31-05-244
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 400 mg Aripiprazole IM Depot (Experimental): 400 mg aripiprazole IM (intramuscular) depot intramuscular injection once every 4 weeks for 5 months. All participants were on a stable dose of 10 mg aripiprazole tablets once daily in the morning for at least 14 days prior to randomization and continued 10 mg aripiprazole tablets once daily on days 1 to 14.
  Interventions: Drug: aripiprazole IM depot; Drug: aripiprazole tablets
- 300 mg Aripiprazole IM Depot (Experimental): 300 mg aripiprazole IM depot intramuscular injection once every 4 weeks for 5 months. All participants were on a stable dose of 10 mg aripiprazole tablets once daily in the morning for at least 14 days prior to randomization and continued 10 mg aripiprazole tablets once daily on days 1 to 14.
  Interventions: Drug: aripiprazole IM depot; Drug: aripiprazole tablets
- 200 mg Aripiprazole IM depot (Experimental): 200 mg aripiprazole IM depot intramuscular injection once every 4 weeks for 5 months. All participants were on a stable dose of 10 mg aripiprazole tablets once daily in the morning for at least 14 days prior to randomization and continued 10 mg aripiprazole tablets once daily on days 1 to 14.
  Interventions: Drug: aripiprazole IM depot; Drug: aripiprazole tablets

INTERVENTIONS:
Drug: aripiprazole IM depot — Aripiprazole IM depot supplied as 200 mg or 400 mg vials of lyophilized aripiprazole powder to prepare for IM injection.
Drug: aripiprazole tablets — Aripiprazole tablets 10 mg once daily in the morning for 14 days.

SUMMARY:
This study will evaluate the safety, tolerability, efficacy and pharmacokinetics of aripiprazole intramuscular (IM) depot multiple doses every 4 weeks in adult patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria
* good physical health as determined by normal medical history, clinical laboratory results, electrocardiograms (ECGs) and physical examinations
* ability to provide informed consent and/or consent from a legally acceptable representation
* body mass index (BMI) of 18 to 35 kg/m^2

Exclusion Criteria:

* sexually active males and females of child-bearing potential who are not practicing double barrier birth control or are not abstinent during the study plus 30 days for female or 90 days for males following the last dose of medication
* history of drug or alcohol abuse within 6 months and/or positive urine drug screen
* participants who consume alcohol beverages routinely
* participants who consume alcohol beverages during the screening period
* use of any antipsychotic medication, other prohibited psychotropic medication, and any cytochrome P450 2D6 (CYP2D6) and cytochrome P450 3A4 (CYP3A4) inhibitors or CYP3A4 inducers within 14 days
* use of any prescription medication unless approved by Medical Monitor or Study Director
* history of current hepatitis or carrier of HBsAg (Hepatitis B surface antigen) and/or Hepatitis C Virus antibodies (anti-HCV)
* females who are pregnant or lactating
* participants who have participated in any clinical trial involving a psychotropic medication within one month prior to enrollment; participants who have participated in a previous IM Depot study within the last 1 year; patients who have previously enrolled and received study medication in an aripiprazole IM Depot clinical trial
* donation of blood or plasma to a blood bank or in a clinical study (except a screening visit)within 30 days prior to enrollment
* any major surgery within 30 days prior to enrollment
* blood transfusion within 30 days prior to enrollment
* evidence of organ dysfunction or any clinically significant deviation from normal in the physical, electrocardiographic, or clinical laboratory examinations
* patient represents a significant risk of committing suicide based on history
* patients currently in an acute relapse
* patients with Axis I (DSM-IV) diagnosis of schizoaffective or bipolar disorder
* patients who are considered treatment-resistant to antipsychotic medication
* patients with a history of neuroleptic malignant syndrome
* any other sound medical reason as determined by the clinical investigator

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Otsuka Investigative Site, Cerritos, California
  - Otsuka Investigative Site, Garden Grove, California
  - Otsuka Investigative Site, Glendale, California
  - Otsuka Investigative Site, Paramount, California
  - Otsuka Investigative Site, St Louis, Missouri
  - Otsuka Investigative Site, Willingboro, New Jersey
  - Otsuka Investigative Site, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Started | 14 | 16 | 11
Safety Population; Received Study Drug | 14 | 15 | 10
Completed | 10 | 8 | 4
Not Completed | 4 | 8 | 7
Not completed — Adverse Event | 0 | 4 | 1
Not completed — Subject met withdrawal criteria | 3 | 2 | 0
Not completed — Subject withdrawn by Investigator | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 5
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot | Total
Number analyzed (Participants) | 14 | 16 | 11 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (9.2) | 43.3 (9.6) | 46.0 (12.7) | 45.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 1 | 12
  Male | 7 | 12 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: Safety and tolerability was assessed by the number of participants with adverse events (AE). An AE was defined as any new medical problem, or exacerbation of an existing problem, experienced by a subject while enrolled in the study, whether or not it was considered drug-related by the investigator. Abnormal laboratory test findings were considered AEs if, in the opinion of the investigator, they represented an abnormal (ie, clinically significant) change from baseline for that individual participant.
Time Frame: 7 Months
Population: Participants who received at least one dose of study medication are included in the safety analysis set.
Measure: Number; unit: Participants
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 14 | 15 | 10
Participants | 11 | 11 | 6

2. Primary Outcome: Aripiprazole Maximum Steady State Plasma Concentration (Css,Max)
Description: Blood samples were collected for pharmacokinetic parameters pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 264, 336, 504, 672, 1008 and 1344 hours post-dose and were analyzed for aripiprazole. Values for Css,max were determined directly from the observed data during the dosing interval (0-1344 hours) after the fifth monthly injection.
Time Frame: Pre-dose and 1 to 1344 hours post-dose at Month 5
Population: Participants who received at least 3 doses of study medication and had pharmacokinetic (pK) samples collected through at least 672 hours following the 5th dose are included in the efficacy pK analysis set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 10 | 8 | 4
ng/mL | 316 (160) | 269 (128) | 100 (68.4)

3. Primary Outcome: Aripiprazole Minimum Steady State Plasma Concentration (Css,Min)
Description: Blood samples were collected for pharmacokinetic parameters pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 264, 336, 504, 672, 1008 and 1344 hours post-dose and were analyzed for aripiprazole. Values for Css,min were determined directly from the observed data at 672 hours after the fifth monthly injection.
Time Frame: 672 hours post-dose at Month 5
Population: Participants who received at least 3 doses of study medication and had pharmacokinetic (pK) samples collected through at least 672 hours following the 5th dose are included in the efficacy pK analysis set. Data was missing for 1 patient in the 200 mg Aripiprazole IM Depot arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 10 | 8 | 3
ng/mL | 212 (113) | 156 (67.7) | 95.0 (86.2)

4. Primary Outcome: Aripiprazole Area Under the Concentration-time Curve at Steady-state (AUCτ)
Description: Blood samples were collected for pharmacokinetic parameters pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 264, 336, 504, 672, 1008 and 1344 hours post-dose and were analyzed for aripiprazole. Values of AUCτ were estimated using the linear trapezoidal rule during each dosing interval from 0 to 1344 hours post-dose.
Time Frame: Pre-dose and 1 to 1344 hours post-dose at Month 5
Population: Participants who received at least 3 doses of study medication and had pharmacokinetic (pK) samples collected through at least 672 hours following the 3rd or 4th dose are included in the efficacy pK analysis set. Data was missing for 1 patient in the 300 mg Aripiprazole IM Depot arm.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 10 | 7 | 4
μg*h/mL | 163 (88.8) | 140 (58.4) | 54.5 (39.4)

5. Secondary Outcome: Aripiprazole Maximum (Peak) Plasma Concentration (Tmax)
Description: Blood samples were collected for pharmacokinetic parameters pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 264, 336, 504, 672, 1008 and 1344 hours post-dose and were analyzed for aripiprazole. Values for tmax were determined directly from the observed data during the dosing interval (0-1344 hours) after the fifth monthly injection.
Time Frame: Pre-dose and 1 to 1344 hours post-dose at Month 5
Population: Participants who received study medication and had pharmacokinetic (pK) samples collected through at least 672 hours following the 5th dose are included in the efficacy pK analysis set.
Measure: Median (Full Range); unit: Day
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 10 | 8 | 4
Day | 7.1 [3.0 to 11.2] | 6.5 [0.5 to 21.2] | 5.0 [4.0 to 27.9]

6. Secondary Outcome: Aripiprazole Steady-state Plasma Concentration (Css,Avg)
Description: Blood samples were collected for pharmacokinetic parameters pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 264, 336, 504, 672, 1008 and 1344 hours post-dose and were analyzed for aripiprazole. Values for Css,avg were determined directly from the observed data during the dosing interval (0-1344 hours) after the fifth monthly injection.
Time Frame: Pre-dose and 1 to 1344 hours post-dose at Month 5
Population: Participants who received study medication and had pharmacokinetic (pK) samples collected through at least 672 hours following the 5th dose are included in the efficacy pK analysis set. Data was missing for 1 patient in the 300 mg Aripiprazole IM Depot arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 10 | 7 | 4
ng/mL | 242 (132) | 208 (87.0) | 81.1 (58.7)

7. Secondary Outcome: Aripiprazole Terminal-phase Elimination Half-life (t1/2,z)
Description: Blood samples were collected for pharmacokinetic parameters pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 264, 336, 504, 672, 1008 and 1344 hours post-dose and were analyzed for aripiprazole. Values for t1/2,z were determined directly from the observed data during the dosing interval (0-1344 hours) after the fifth monthly injection.
Time Frame: Pre-dose and 1 to 1344 hours post-dose at Month 5
Population: Participants who received at least 3 doses of study medication and had pharmacokinetic (pK) samples collected through at least 672 hours following the 3rd or 4th dose are included in the efficacy pK analysis set. The analysis population for this outcome measure represents a sub-set who were evaluable for this measure at month 5.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 6 | 4 | 0
Day | 46.5 (10.8) | 29.9 (8.0) |

8. Secondary Outcome: Dehydro-aripiprazole Maximum Steady State Plasma Concentration (Css,Max)
Description: Blood samples were collected for pharmacokinetic parameters pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 264, 336, 504, 672, 1008 and 1344 hours post-dose and were analyzed for dehydro-aripiprazole. Values for Css,max were determined directly from the observed data during the dosing interval (0-1344 hours) after the fifth monthly injection.
Time Frame: Pre-dose and 1 to 1344 hours post-dose at Month 5
Population: Participants who received at least 3 doses of study medication and had pharmacokinetic (pK) samples collected through at least 672 hours following the 3rd or 4th dose are included in the efficacy pK analysis set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 10 | 8 | 4
ng/mL | 89.4 (37.9) | 74.7 (20.8) | 30.3 (19.8)

9. Secondary Outcome: Dehydro-aripiprazole Minimum Steady State Plasma Concentration (Css,Min)
Description: Blood samples were collected for pharmacokinetic parameters pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 264, 336, 504, 672, 1008 and 1344 hours post-dose and were analyzed for dehydro-aripiprazole. Values for Css,min were determined directly from the observed data during the dosing interval (0-1344 hours) after the fifth monthly injection.
Time Frame: Pre-dose and 1 to 1344 hours post-dose at Month 5
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 10 | 8 | 4
ng/mL | 64.1 (27.0) | 54.1 (21.1) | 26.2 (24.7)

10. Secondary Outcome: Dehydro-aripiprazole Area Under the Concentration-Time Curve at Steady-State (AUCτ)
Description: Blood samples were collected for pharmacokinetic parameters pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 264, 336, 504, 672, 1008 and 1344 hours post-dose and were analyzed for dehydro-aripiprazole. Values of AUCτ were estimated using the linear trapezoidal rule during each dosing interval from 0 to 1344 hours post-dose.
Time Frame: Pre-dose and 1 to 1344 hours post-dose at Month 5
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 10 | 8 | 4
μg*h/mL | 47.8 (19.1) | 38.9 (13.2) | 14.7 (9.47)

11. Secondary Outcome: Dehydro-aripiprazole Maximum (Peak) Plasma Concentration (Tmax)
Description: Blood samples were collected for pharmacokinetic parameters pre-dose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 264, 336, 504, 672, 1008 and 1344 hours post-dose and were analyzed for dehydro-aripiprazole. Values for tmax were determined directly from the observed data during the dosing interval (0-1344 hours) after the fifth monthly injection.
Time Frame: Pre-dose and 1 to 1344 hours post-dose at Month 5
Population: as for outcome 8
Measure: Median (Full Range); unit: Day
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 10 | 8 | 4
Day | 6.6 [3.0 to 14.0] | 12.5 [0.5 to 22.2] | 5.5 [0.0 to 27.9]

12. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at Week 12 and Week 24
Description: The PANSS consisted of 3 subscales with a total of 30 symptom constructs each rated on a 7-point scale where 1=absence of symptoms to 7=extremely severe symptoms. The Positive Subscale consisted of 7 positive symptom constructs with a possible subscale score of 7 to 49, the Negative Subscale consisted of 7 negative symptom constructs with a possible subscale score of 7 to 49 and the General Psychopathology Subscale consisted of 16 symptom constructs for a possible subscale score of 16 to 112. The PANSS Total Score ranged from 30 (best) to 210 (worst; indicating more severe symptoms). A Negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12, Week 24
Population: All randomized participants with data available were included in this analysis population-last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 13 | 14 | 10
units on a scale
  Week 12 | 0.0 (20.2) | 1.1 (12.1) | -1.3 (4.8)
  Week 24 | -0.8 (20.9) | -1.6 (14.1) | -1.3 (5.3)

13. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Positive Subscale Scores at Week 12 and Week 24
Description: The PANSS Positive Subscale consisted of 7 symptom constructs: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. Severity was rated on a 7-point scale where 1=absence of symptoms to 7=extremely severe symptoms. The total score on the Positive Subscale ranged from 7 to 49 with a higher score indicating more severe symptoms. A Negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12, Week 24
Population: All randomized participants with data available were included in this analysis population (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 13 | 14 | 10
units on a scale
  Week 12 | -1.2 (6.1) | 1.3 (4.0) | -1.0 (1.2)
  Week 24 | -1.6 (6.1) | 0.4 (4.5) | -1.0 (1.6)

14. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Negative Subscale Scores at Week 12 and Week 24
Description: The PANSS Negative Subscale consisted of 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. Severity was rated on a 7-point scale where 1=absence of symptoms to 7=extremely severe symptoms. The total score on the Negative Subscale ranged from 7 to 49 with a higher score indicating more severe symptoms. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12, Week 24
Population: All randomized participants with data available were included in this analysis population (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 13 | 14 | 10
units on a scale
  Week 12 | 1.1 (4.4) | 0.1 (3.2) | 0.0 (2.0)
  Week 24 | 0.5 (4.2) | -0.1 (3.7) | -0.6 (2.0)

15. Secondary Outcome: Change From Baseline in the Clinical Global Impression- Severity of Illness Score (CGI-S) at Week 12 and Week 24
Description: The severity of illness for each participant was rated using the CGI-S scale. The investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" using an 8-point scale where 0=not assessed to 7=among the most extremely ill patients. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12, Week 24
Population: All randomized participants with data available were included in this analysis population (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 14 | 16 | 10
units on a scale
  Week 12 | -0.1 (0.5) | 0.0 (0.6) | -0.2 (0.4)
  Week 24 | -0.1 (0.5) | -0.1 (0.7) | -0.2 (0.4)

16. Secondary Outcome: Clinical Global Impression-Improvement Scale (CGI-I) at Week 12 and Week 24
Description: The participant's overall improvement was rated for each participant using the CGI-I scale. The investigator rated the participant's total improvement by answering the following question: "Compared to his/her condition at baseline (prior to randomization), how much has the patient changed?" using an 8-point scale where 0=not assessed, 1=very much improved to 7=very much worse. Lower scores indicated improvement.
Time Frame: Baseline, Week 12, Week 24
Population: All randomized participants with data available at the given time-point were included in this analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 13 | 15 | 9
units on a scale
  Week 12 (n=12, 13, 9) | 3.3 (0.9) | 3.6 (0.8) | 3.4 (0.7)
  Week 24 | 3.7 (1.0) | 3.4 (0.7) | 3.7 (0.7)

17. Secondary Outcome: Number of Participants Hospitalized for Adverse Event "Worsening Schizophrenia"
Description: The number of participants hospitalized for the Adverse Event "Worsening Schizophrenia included all participants who were hospitalized for any Adverse Event pertaining to the exacerbation of schizophrenic symptoms.
Time Frame: 7 Months
Population: All randomized participants were included in the analysis population.
Measure: Number; unit: Participants
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Number analyzed (Participants) | 14 | 16 | 11
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Description: Safety Population included all randomized participants who received study drug.
Arm/Group | 400 mg Aripiprazole IM Depot | 300 mg Aripiprazole IM Depot | 200 mg Aripiprazole IM Depot
Serious Adverse Events (participants affected / at risk) | 0/14 | 3/15 | 0/10
Other Adverse Events (participants affected / at risk) | 9/14 | 10/15 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 mg Aripiprazole IM Depot (N=14) | 300 mg Aripiprazole IM Depot (N=15) | 200 mg Aripiprazole IM Depot (N=10)
Chest Pain (General disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 400 mg Aripiprazole IM Depot (N=14) | 300 mg Aripiprazole IM Depot (N=15) | 200 mg Aripiprazole IM Depot (N=10)
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Cyst (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1
Injection site discomfort (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 4 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Bed bug infestation (Infections and infestations) | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Infected insect bite (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood magnesium increased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 2 | 1
Glucose urine present (Investigations) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Akathisia (Nervous system disorders) | 1 | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1 | 0
Dystonia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 2
Sedation (Nervous system disorders) | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 1
Tremor (Nervous system disorders) | 3 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Drug dependence (Psychiatric disorders) | 0 | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1
Nightmare (Psychiatric disorders) | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No